CLINICAL TRIAL: NCT05214430
Title: Exclusive Enteral Nutrition for Remissionof Crohn's Diseases After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Weiming, Jinling Hospital, China, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: jinlingH202001
Record Dates: First submitted 2022-01-26; First posted 2022-01-28 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease in Remission

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 months exclusive enteral nutrition after surgery (Experimental): 3 months exclusive enteral nutrition after surgery
  Interventions: Other: 3 months exclusive enteral nutrition after surgery
- less than 1 months exclusive enteral nutrition after surgery (Experimental): less than 1 months exclusive enteral nutrition after surgery
  Interventions: Other: 3 months exclusive enteral nutrition after surgery

INTERVENTIONS:
Other: 3 months exclusive enteral nutrition after surgery — patients underwent intestinal resection and anastomosis in this arm will given over 3 months exclusive enteral nutrition,and free diet after 3 months.

SUMMARY:
For patients with Crohn's diseases undergoing surgery，whether postoperative exclusive enteral nutrition(EEN) could delay the endoscopic relapse needs exploration.The trial will investigate the efficacy of postoperative EEN for maintaining disease remission.

ELIGIBILITY:
Inclusion Criteria:

- CD patients who undergoing bowel resection with anastomosis

Exclusion Criteria:

* patients who received stoma creation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
postoperative endoscopic recurrence | 1 YEAR
  over i2b of rutgeerts score

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Institute,Jinling Hospital,Nanjing,Jiangsu,China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duan M, Lu M, Diao Y, Cao L, Wu Q, Liu Y, Gong J, Zhu W, Li Y. Azathioprine Plus Exclusive Enteral Nutrition Versus Azathioprine Monotherapy for the Prevention of Postoperative Recurrence in Patients with Crohn's Disease: An Open-Label, Single-Centre, Randomized Controlled Trial. J Crohns Colitis. 2024 Aug 6;18(7):1113-1121. doi: 10.1093/ecco-jcc/jjae015. PMID 38253914